CLINICAL TRIAL: NCT01495455
Title: Nottingham Osteoarthritis Biomarker Study 2011
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 11049
Record Dates: First submitted 2011-11-30; First posted 2011-12-20 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, urine and synovial fluid.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Knee osteoarthritis
- No knee pain/osteoarthritis

SUMMARY:
Osteoarthritis is by far the most common joint condition and the single largest cause of disability in the older population. The investigators still have a poor understanding of the nature of osteoarthritis and factors that influence its development and progression. Identification of biochemical markers that relate to cartilage loss, bony overgrowth and other features that occur with osteoarthritis will advance our understanding. Over the last 5 years analytical methods have developed to measure a range of different biomarkers. This pilot study will use these analytical methods to measure biomarker levels in joint fluid, urine and blood of 50 participants with Osteoarthritis (OA) and 50 healthy volunteers.

This study will provide novel pilot data on the changes in the composition of the synovial fluid, urine and blood in patients with OA. Apart from being a key target site for OA, the knee is a suitable joint for study because of its accessibility to clinical assessment, joint aspiration and imaging.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* Be able to provide written informed consent
* Aged 30 and over

Knee OA patients:

• Radiographic signs of OA - that is definite joint space narrowing plus osteophyte in at least one compartment of the knee

Normal controls:

* No knee pain
* No clinical or radiographic changes of knee OA

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Secondary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Difference in the levels of pro-inflammatory and anti-inflammatory lipids mediators between individuals with knee osteoarthritis and those with normal knees. | within 6 months of recruitment of last participant

CONTACTS AND LOCATIONS:
Overall Officials: Michael Doherty, MA MB FRCP, Principal Investigator — University of Nottingham
Locations (1):
- Academic Rheumatology, University of Nottingham, Nottingham, United Kingdom